CLINICAL TRIAL: NCT00424411
Title: Efficacy and Safety of Inhaled Compared With Subcutaneous Human Insulin Therapy in Subjects With Type 2 Diabetes Mellitus: A Six-Month, Outpatient, Parallel Comparative Trial
Brief Title: Six Month Clinical Trial Assessing Efficacy And Safety Of Inhaled Insulin In Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 217-108
Record Dates: First submitted 2007-01-17; First posted 2007-01-19 (Estimated); Last update posted 2007-02-13 (Estimated); Status verified 2007-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exubera

INTERVENTIONS:
Drug: Inhaled human insulin (EXUBERA™)

SUMMARY:
To determine, in subjects with Type 2 Diabetes Mellitus:

1. Whether glycemic control can be achieved at least as effectively with an insulin regimen involving pre-meal EXUBERA™ (inhaled insulin) plus a single bedtime Ultralente injection as with a conventional subcutaneous insulin regimen involving 2 mixed Regular/NPH insulin injections per day.
2. The toleration and safety of EXUBERA™ (inhaled insulin) therapy and its effects after 6 months, if any, on measures of pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* Stable insulin regimen of at least 2 injections per day

Exclusion Criteria:

* Any smoking within the last 6 months. Smoking is not permitted at any time during this study.
* Subjects on insulin pump during 2 months prior to screening.
* Subjects with poorly-controlled asthma, clinically significant chronic obstructive pulmonary disease, or other significant respiratory disease.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 1999-09; Study Completion 2000-12

PRIMARY OUTCOMES:
Primary outcome is 24 week change in baseline in HbA1c.

SECONDARY OUTCOMES:
The secondary endpoints include the following efficacy assessments:
Incidence of hypoglycemia
Proportion of subjects with acceptable glycemic control (e.g., HbA1c<8%)
Change from baseline in fasting lipid profile
Change from baseline in fasting plasma glucose level
Change from baseline in meal glucose response (2-hour postprandial increment in plasma glucose)
Dose of insulin (total dose of injected sustained-duration insulin, and total dose of inhaled or injected Regular insulin during the study).
Change from baseline in body weight
Change from baseline in 24-hour home glucose profile (based on the area under the glucose profile curve calculated by the trapezoid rule with special weights assigned to the pre-breakfast and bedtime assessments).
Patient satisfaction and preference.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (45):
- United States (34):
  - Pfizer Investigational Site, Burlingame, California
  - Pfizer Investigational Site, Irvine, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, New Hyde Park, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Greenville, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Irving, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Burlington, Vermont
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Renton, Washington
- Canada (11):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Red Deer, Alberta
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, St. John's, Newfoundland and Labrador
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Mississauga, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Chomedy, Quebec
  - Pfizer Investigational Site, Montreal, Quebec

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=108&StudyName=Six+Month+Clinical+Trial+Assessing+Efficacy+And+Safety+Of+Inhaled+Insulin+In+Type+2+Diabetes